CLINICAL TRIAL: NCT01934283
Title: Intrabdominal Pressure in Small Bowel Obstruction as a Possible Predictor for the Need of Operation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Meir Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: mmc-0188-12
Record Dates: First submitted 2013-02-27; First posted 2013-09-04 (Estimated); Last update posted 2013-09-04 (Estimated); Status verified 2013-08

CONDITIONS: Small Bowel Obstruction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- operated patients (No Intervention): small bowel obstrucion patients who needed surgery for treatment of obstruction.
  Interventions: Device: urine folly catheter

INTERVENTIONS:
Device: urine folly catheter

SUMMARY:
Small bowel obstruction (SBO) is a common surgical diagnosis. Most of SBO are related to post operative adhesions and most of them resolve without the need of surgical intervention. The most important thing dealing with SBO is to identify the more complex obstructions that need surgery.

Some clinical, physiological and radiological signs are recognized as markers of a more complex obstruction.

The pathophysiology of bowel obstruction is explained as damage created by pressure on the abdominal wall causing ischemia. Yet there are no studies, as far as we know, that measure intra-abdominal pressure in SBO patients and it relation to the severity of the obstruction.

In this study we will measure the intra-abdominal pressure in SBO patients systematically and we will examine if more severe obstructions are accompanied by elevated intra-abdominal pressure.

ELIGIBILITY:
Inclusion Criteria:

* older than 18 , diagnosis of small bowel obstruction

Exclusion Criteria:

* younger then 18 , pregnant women, large bowel obstruction, incarcerated hernia, large ventral hernia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 125 (Estimated)
Dates: Start 2013-10; Primary Completion 2015-06 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
intra abdominal pressure | up to 1 week
  serial intraabdominal pressure will be measured during hospitalisation up to discharge or operation.

CONTACTS AND LOCATIONS:
Locations (1):
- Meir Medical Center, Kfar Saba, Israel